CLINICAL TRIAL: NCT02947984
Title: Prospective Study Of Patients With Recurrent Or Incomplete Excised Benign Intercranial Meningiomas For The Evaluation Of Treatment Result With Combined Proton And Photon Irradiation To Doses 55.8 Or 63.0 CGE
Brief Title: Proton/Photon Rt - Benign Meningiomas(P92-13)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Helen A. Shih, MD, Prinicipal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97-550
Record Dates: First submitted 2007-12-28; First posted 2016-10-28 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Benign Meningioma
Keywords: sphenoid region; parasellar area; photon radiation therapy; proton radiation therapy
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment (Experimental): Standard radiation therapy: 55.8 CGE in 31 treatments of 1.8 CGE given once a day, for five days each week.
  Interventions: Radiation: Standard Treatment
- Higher Dose Treatment (Experimental): 63 CGE in 35 treatments of 1.8 CGE given once a day, for five days of each week.
  Interventions: Radiation: Higher Dose

INTERVENTIONS:
Radiation: Standard Treatment — 55.8 CGE in 31 treatments of 1.8 CGE given once a day, for five days each week. Treatment based upon a treatment planning CT.
  Arms: Standard Treatment
Radiation: Higher Dose — 55.8 CGE in 31 treatments of 1.8 CGE given once a day, for five days each week. Treatment based upon a treatment planning CT.
  Arms: Higher Dose Treatment

SUMMARY:
The purpose of this study is to determine the best radiation dose for participants with meningioma that has grown back after previous surgery, or which the surgeon has been unable to remove completely. This research study is designed to determine whether a higher dose of radiation will decrease the likelihood that the tumor will grow back, compared to the probability of re-growth that occurs after standard radiation doses.

DETAILED DESCRIPTION:
* After initial interview and physical examination, an immobilization device (head mask, neck support, back support, etc.) will be made for the participant. A treatment planning CT will be performed and a radiation treatment plan will be based on this CT scan.
* The radiation dose will usually be given once a day, five days per week. The radiation treatment will take between 7 and 8 1/2 weeks, including treatment planning.
* Treatment doses will vary, and the dose each participant will receive will be made on the basis of random assignment. Participants will either receive the usual dose of 55.8 CGE in 31 treatments or 1.8 CGE, or 63 CGE in 35 treatments of 1.8 CGE.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Histological documentation of benign meningioma
* Documentation by imaging studies (CT and/ or MRI) or residual or recurrent intracranial tumor
* Karnofsky performance status of ≥ 70
* Study specific informed consent

Exclusion Criteria:

* Malignant meningiomas
* Prior cranial irradiation, except treatment of localized skin cancer of the face or scalp
* Patients having a concurrent primary cancer (except skin)
* Patients having another cancer controlled < 3 years
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 1999-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen A Shih, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hosital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment: Standard radiation therapy: 55.8 CGE in 31 treatments of 1.8 CGE given once a day, for five days each week.
  Standard Treatment: 55.8 CGE in 31 treatments of 1.8 CGE given once a day, for five days each week.
  Treatment based upon a treatment planning CT.
Period: Overall Study
Arm/Group | Standard Treatment | Higher Dose Treatment
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Higher Dose Treatment | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Median (Full Range); unit: years] | 61 [31 to 77] | 50.5 [38 to 76] | 55.5 [31 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44
Tumor Location [Number; unit: Tumors] — Count of tumors by location
  Tumors
    Sphenoid wing | 7 | 8 | 15
    Cavernous sinus | 3 | 8 | 11
    Sella/Parasella | 6 | 2 | 8
    Cerebellar pontine angle | 3 | 1 | 4
    Clival/prepontine space | 3 | 1 | 4
    Olfactory groove | 1 | 0 | 1
    Optic canal | 0 | 1 | 1
    Tentorium | 0 | 1 | 1
Smoking Status [Count of Participants; unit: Participants]
  Smoker | 9 | 13 | 22
  Non-smoker | 11 | 6 | 17
  Unknown | 2 | 3 | 5
Co-morbidities [Number; unit: participants]
  Hypertension | 3 | 6 | 9
  Diabetes mellitus | 0 | 4 | 4
  Hyperlipidemia | 1 | 0 | 1
  Coronary artery disease | 1 | 0 | 1
  One or more of the above | 4 | 6 | 10
Radiation Indication [Count of Participants; unit: Participants]
  Sub-Total Resection, postoperative | 11 | 12 | 23
  Recurrent Disease | 11 | 10 | 21
Gross Tumor Volume [Median (Full Range); unit: Cubic Centimeters] | 39.7 [5.6 to 243] | 13.2 [3 to 313] | 26.5 [3 to 313]
Clinical Target Volume [Median (Full Range); unit: Cubic Centimeters] | 49 [9 to 464] | 28 [6.5 to 150.7] | 38.5 [6.5 to 464]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The number of participants surviving at the given time point. Progression free survival (PFS) is measured from the starting date of radiation therapy and analyzed by intention to treat. PFS is measured until the earlier, date of death or development of radiologic progression, and is otherwise censored at the last follow-up for progression-free patients still alive.
Time Frame: 5, 10, 15 years
Population: Progression free survival in the entire cohort and by radiation indication sub-groups
Measure: Number (95% Confidence Interval); unit: percentage of participants surviving
Arm/Group | Standard Treatment | Higher Dose Treatment
Number analyzed (Participants) | 22 | 22
percentage of participants surviving
  Entire Cohort: 5 Years | 91 [68 to 98] | 91 [68 to 98]
  Entire Cohort: 10 Years | 86 [62 to 95] | 81 [58 to 93]
  Entire Cohort: 15 Years | 52 [28 to 72] | 70 [45 to 86]
  Subtotal Resection: 5 Years: number analyzed (Participants) | 11 | 12
  Subtotal Resection: 5 Years | 100 [NA to NA] — confidence interval not defined because no deaths occurred | 83 [48 to 96]
  Subtotal Resection: 10 Years: number analyzed (Participants) | 11 | 12
  Subtotal Resection: 10 Years | 91 [51 to 99] | 67 [34 to 86]
  Subtotal Resection: 15 Years: number analyzed (Participants) | 11 | 12
  Subtotal Resection: 15 Years | 64 [30 to 85] | 57 [25 to 80]
  Recurrent Disease: 5 Years: number analyzed (Participants) | 11 | 10
  Recurrent Disease: 5 Years | 82 [45 to 95] | 100 [NA to NA] — confidence interval not defined because no deaths occurred
  Recurrent Disease: 10 Years: number analyzed (Participants) | 11 | 10
  Recurrent Disease: 10 Years | 82 [45 to 95] | 100 [NA to NA] — confidence interval not defined because no deaths occurred
  Recurrent Disease: 15 Years: number analyzed (Participants) | 11 | 10
  Recurrent Disease: 15 Years | 65 [24 to 88] | 100 [NA to NA] — confidence interval not defined because no deaths occurred
Statistical Analysis 1: Comparison: Standard Treatment vs Higher Dose Treatment; Null hypothesis: Progression free survival is not significantly different by dose level in the overall cohort; Test type: Other; p = 0.234, Log Rank
Statistical Analysis 2: Comparison: Standard Treatment vs Higher Dose Treatment; Null hypothesis: Progression free survival is not significantly different by dose level in the subgroup receiving treatment due to a sub-total resection; Test type: Other; p = .820, Log Rank
Statistical Analysis 3: Comparison: Standard Treatment vs Higher Dose Treatment; Null hypothesis: Progression free survival is not significantly different by dose level in the sub-group receiving treatment due to recurrent disease; Test type: Other; p = .061, Log Rank

2. Secondary Outcome: Acute Toxicities
Description: The number of participants that experienced the specified acute toxicities (any grade) as assessed by Radiation Therapy Oncology Acute Morbidity Scoring Criteria. Acute toxicities were assessed from the start of treatment through day 90 of treatment.
Time Frame: 90 Days
Measure: Number; unit: participants
Arm/Group | Standard Treatment | Higher Dose Treatment
Number analyzed (Participants) | 22 | 22
participants
  Vision loss | 2 | 1
  Visual field deficit | 1 | 0
  Diplopia | 2 | 0
  Ptosis | 0 | 1
  Exophthalmos | 1 | 0
  Conjunctivitis | 1 | 2
  Eye, other | 2 | 5
  Hearing loss | 1 | 2
  Tinnitus | 0 | 1
  Olfactory alteration | 1 | 1
  Gustation alteration | 3 | 1
  Neuromotor deficit | 1 | 0
  Weakness | 1 | 0
  Facial numbness | 2 | 1
  Facial weakness | 2 | 2
  Ataxia | 1 | 0
  Seizure | 1 | 1
  Headache | 3 | 8
  Nausea | 9 | 8
  Dizziness | 1 | 1
  Vertigo | 1 | 4
  Syncope | 1 | 0
  Depression | 0 | 3
  Neurocog deficit | 1 | 3
  Endocrine deficit | 0 | 1
  Skin changes | 16 | 18
  Alopecia | 7 | 11
  Fatigue | 12 | 10

3. Secondary Outcome: Late Toxicities
Description: The number of participants that experienced the specified late toxicities (any grade) as assessed by Radiation Therapy Oncology Group Late Effects Scale.
Time Frame: 5 Years
Measure: Number; unit: participants
Arm/Group | Standard Treatment | Higher Dose Treatment
Number analyzed (Participants) | 22 | 22
participants
  Vision loss | 5 | 2
  Visual field deficit | 5 | 1
  Diplopia | 1 | 3
  Exophthalmos | 0 | 2
  Eye, other | 3 | 2
  Hearing loss | 6 | 4
  Tinnitus | 2 | 3
  Olfactory alteration | 0 | 2
  Gustation alteration | 0 | 1
  Dysphasia | 0 | 1
  Neuromotor deficit | 1 | 0
  Weakness | 1 | 2
  Facial numbness | 1 | 4
  Facial weakness | 4 | 2
  Ataxia | 2 | 3
  Fall | 0 | 3
  Dysarthria | 1 | 0
  Headache | 5 | 3
  Dizziness | 1 | 0
  Vertigo | 1 | 1
  Depression | 0 | 1
  Neurocognative deficit | 7 | 6
  Endocrine deficit | 7 | 10
  Osteoporosis | 0 | 1
  Cerebral edema | 1 | 0
  Brain atrophy | 0 | 1
  Skin changes | 1 | 1
  Alopecia | 0 | 2
  Fatigue | 4 | 3

4. Secondary Outcome: Local Failure Rate
Description: The number of participants with local failure. Local failure is defined as radiologic progression seen on follow-up scans showing tumor margin(s) extending in any direction at least five mm beyond that seen on baseline scans.
Time Frame: 15 Years
Population: Failure rates are shown by dose group in the overall study population and by treatment indication subgroups.
Measure: Number; unit: participants
Arm/Group | Standard Treatment | Higher Dose Treatment
Number analyzed (Participants) | 22 | 22
participants
  Entire Cohort | 3 | 2
  Post-operative subgroup: number analyzed (Participants) | 11 | 12
  Post-operative subgroup | 0 | 1
  Tumor recurrence subgroup: number analyzed (Participants) | 11 | 10
  Tumor recurrence subgroup | 3 | 1

ADVERSE EVENTS:
Time Frame: 90 Days, 15 years
Description: Patients were assessed for adverse events with Radiation Therapy Oncology Group Common Toxicity Criteria. Patients were assessed weekly during the course of treatment. Post treatment, participants were evaluated for interval history and neurological function routinely at one month, every three months during the first year, four month intervals during the second year, twice yearly through year 5, and then yearly for the remainder of follow-up.
Arm/Group | Standard Treatment | Higher Dose Treatment
All-Cause Mortality (participants affected / at risk) | 14/22 | 5/22
Serious Adverse Events (participants affected / at risk) | 6/22 | 0/22
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Treatment (N=22) | Higher Dose Treatment (N=22)
Neuromotor deficit (Nervous system disorders) | 2 | 0
Vision loss (Eye disorders) | 2 | 0
Endocrine deficit (Endocrine disorders) | 1 | 0
Cerebral edema (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Treatment (N=22) | Higher Dose Treatment (N=22)
Vision loss (Eye disorders) | 5 | 3
Visual field deficit (Eye disorders) | 6 | 1
Diplopia (Eye disorders) | 3 | 3
Ptosis (Eye disorders) | 0 | 1
Exophthalmos (Eye disorders) | 1 | 2
Conjunctivitis (Eye disorders) | 1 | 2
Eye, other (Eye disorders) | 5 | 7
Hearing loss (Ear and labyrinth disorders) | 7 | 6
Tinnitus (Ear and labyrinth disorders) | 2 | 4
Olfactory alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Gustation alteration (Gastrointestinal disorders) | 3 | 2
Dysphasia (Gastrointestinal disorders) | 0 | 1
Neuromotor deficit (Nervous system disorders) | 0 | 0
Weakness (General disorders) | 2 | 2
Facial numbness (Nervous system disorders) | 3 | 5
Facial weakness (Musculoskeletal and connective tissue disorders) | 6 | 4
Ataxia (Nervous system disorders) | 3 | 3
Fall (General disorders) | 0 | 3
Seizure (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 8 | 11
Nausea (Gastrointestinal disorders) | 9 | 8
Dizziness (Nervous system disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 5
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 4
Neurocog deficit (Nervous system disorders) | 8 | 9
Endocrine deficit (Endocrine disorders) | 6 | 11
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral edema (Nervous system disorders) | 0 | 0
Brain atrophy (Nervous system disorders) | 0 | 1
Skin changes (Skin and subcutaneous tissue disorders) | 17 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 13
Fatigue (General disorders) | 16 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes